CLINICAL TRIAL: NCT02539004
Title: Ultrasound Non-contrast Computed Tomography Real-time Fusion for Urinary Stones Follow up
Brief Title: US-Non Contrast Computed Tomography Real-time Fusion for Urinary Stones Follow up
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0117-15
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Urolithiasis; Ureterolithiasis
Keywords: kidney stones; ureteral stones
MeSH Terms: conditions — Urolithiasis; Ureterolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ultrasound study — Ultrasound study using real-time image fusion with a previous NCCT

SUMMARY:
Urolithiasis is a universal problem, a large part of patients will be affected by multiple stones throughout their lifetime, with estimated recurrence rates of 75% within 20 years. The high recurrence rate requires an increasing amount of imaging follow-up. US-NCCT real-time fusion (Fusion) enables lesion assessment and follow up using both modalities as reference for each other. Our study proposes a novel approach for short term follow up of patients using Fusion instead of repeat NCCT exams.

the goal of the study is to create an initial proof of concept that Fusion is effective for follow up of known urinary stones.

the study is a prospective study on Patients with an obstructing ureteral stone found on a NCCT. Patients will undergo Fusion (using General Electric Logiq E9) after NCCT. The primary endpoint was the ability to locate the ureteral stone using US with guidance of the NCCT as a "Road Map".

ELIGIBILITY:
Inclusion Criteria:

* NCCT within 3 months prior to the US study with proved Urolithiasis

Exclusion Criteria:

* Inability to perform a US study.
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with proved urolithiasis on NCCT
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-06; Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
US identification of ureteral stone seen on NCCT | up to 3 months after NCCT

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Bercovich, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Haifa, Select A State, Israel